CLINICAL TRIAL: NCT03716635
Title: Effect of Intracanal Cryotherapy on Postoperative Pain in Molar Teeth With Symptomatic Irreversible Pulpitis and Apical Periodontitis
Brief Title: Effect of Cryotherapy on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magy Essam Sayed El-Askary, resident at endodontic department cairo university, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-10-19
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Cryotherapy; Saline Solution

STUDY DESIGN:
Intervention Model Description: A random sequence will be generated by computer software, (http://www.random.org/).
  The table will be kept with the assistant supervisor.
Who Masked: Participant
Masking Description: After determining the eligibility of the patient, the assistant supervisor will be contacted to assign the participant to either the intervention (cryotherapy) or the control (normal saline) groups according to the random sequence generated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryotherapy (Experimental): 2.5c cold saline as a final flush after chemicomechanical debridement
  Interventions: Procedure: cryotherapy
- normal saline (Other): room temperature saline is used as a final flush after chemicomechanical preparation
  Interventions: Procedure: normal saline

INTERVENTIONS:
Procedure: cryotherapy — 2.5c cold saline is used as a final flush after chemomechanical preparation
  Arms: cryotherapy
Procedure: normal saline — a room temperature saline is used as a final flush after mechanical preparation
  Arms: normal saline

SUMMARY:
the aim of the study is to evaluate the effect of cryotherapy on postoperative pain in molar teeth with irreversible pulpitis and apical periodontitis

DETAILED DESCRIPTION:
the purpose of the study was to evaluate the effect of 2.5c cold saline irrigation as a final irrigant on postoperative pain after single visit root canal treatment of teeth with vital pulp and apical periodontitis .thirty patients will be included in the study .the teeth will be divided into 2 groups (i.e the control group and the cryotherapy group ) in the cryotherapy group ,final irrigation with 2.5c cold saline solution for 5 mins will be performed following completion of biomechanical preparation whereas in control group same solution stored at room temperature will be used . treatment will be done in a single visit then participants will be asked to rate the intensity of postoperative pain using numerical rating scale at 6,12,24,48 hrs

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years old.
* Systemically healthy patient (ASA I or II).
* mandibular first molar teeth with:
* Preoperative sharp pain and Symptomatic apical periodontitis .absence or slight widening in the periodontal ligament (PDL). .Vital response of pulp tissue to cold pulp tester (ethyl chloride spray).
* Ability for isolation with rubberdam.
* Restorable teeth
* Ability to fill the root canals in single visit treatment.

Exclusion Criteria:

* Teeth without good apical constriction, such as wide or open apex
* Use of any type of analgesics or antibiotic medications within 3 days .Pregnant or nursing females.
* Patients having significant systemic disorder (ASA III or IV).
* Teeth that have :

Non vital pulp tissues. Association with swelling or fistulous tract Acute or chronic periapical abscess Greater than grade I mobility Pocket depth greater than 5 mm No possible restorability

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
postoperative pain assessed by NRS | up to 48 hrs postoperative pain
  Primary outcome (post-operative pain) will be collected by the operator through (NRS) which is an 11 point scale consisting of numbers from 0 through 10 0: reading represents "no pain"
  1- 3: readings represent "mild pain" 4- 6: readings represent "moderate pain" 7- 10: readings represent "severe pain"

SECONDARY OUTCOMES:
amount of analgesics assessed by counting | up to 48 hrs postoperatively
  number of analgesics tablets up to 48 hrs postoperatively

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gundogdu EC, Arslan H. Effects of Various Cryotherapy Applications on Postoperative Pain in Molar Teeth with Symptomatic Apical Periodontitis: A Preliminary Randomized Prospective Clinical Trial. J Endod. 2018 Mar;44(3):349-354. doi: 10.1016/j.joen.2017.11.002. Epub 2018 Feb 3. PMID 29398090